CLINICAL TRIAL: NCT03442452
Title: A Pilot Feasibility and Preliminary Efficacy Study of an Electronic Decision Aid for Patients With Acute Myeloid Leukemia (AML)
Brief Title: AML Electronic Decision Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00091220
Record Dates: First submitted 2018-02-02; First posted 2018-02-22 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-03

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: For this study, we will test the feasibility and preliminary efficacy of utilizing a novel electronic decision aid to improve AML patients' understanding of their illness, prognosis, and treatment options.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electronic Decision Aid (Other): For this study, we will be testing a novel electronic decision aid to improve Acute Myeloid Leukemia patients' understanding of their illness, prognosis, and treatment options.
  Interventions: Other: Electronic Decision Aid Tool

INTERVENTIONS:
Other: Electronic Decision Aid Tool — The AML Decision Aid tool consists of ten video modules, approximately 3 minutes each, containing content regarding key areas such as an explanation of what AML is, treatment choices, and things to consider when determining a treatment path.

SUMMARY:
The purpose of this study is to test the feasibility and preliminary efficacy of a novel electronic decision aid to improve AML patients' understanding of their illness, prognosis, and treatment options.

DETAILED DESCRIPTION:
The purpose of this study is to test the feasibility and preliminary efficacy of a novel electronic decision aid to improve AML patients' understanding of their illness, prognosis, and treatment options. The objective of our program of research is to ultimately improve understanding about what patients with Acute Myeloid Leukemia (AML) know and understand about their disease, as well as what kind of information AML patients want or need to further inform them about the treatment decisions they face.

The AML Decision Aid tool consists of ten video modules, approximately 3 minutes each, containing content regarding key areas such as an explanation of what AML is, treatment choices, and things to consider when determining a treatment path. Recruited subjects will complete a series of surveys, both before viewing of the videos and after

ELIGIBILITY:
Inclusion Criteria:

* At least age 18
* Capacity to give consent
* Diagnosis of acute myeloid leukemia (AML)
* Fluent in English
* Receiving care at Duke, and fits into one of the following scenarios:

  * has not yet made a treatment decision (in the DCI clinics or on the inpatient wards),
  * have recently made a decision (in the last 6 weeks), and are admitted for chemotherapy on 9100 or in the oncology treatment center to receive outpatient therapy,
  * or, during remission, while receiving consolidation chemotherapy in the hospital

Exclusion Criteria:

* Patients too sick to participate per clinician discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Number of enrolled subjects who have completed the study | 1 day
  Feasibility will be determined by enrolled subjects who complete the study (including watching all videos, and completing the surveys).

SECONDARY OUTCOMES:
Change in knowledge about AML after video viewing | Day 1. Pre-video screening and post-video
  Efficacy will be measured by change in knowledge about AML, (including knowledge about the disease itself, and comprehending AML treatment choices and their risks, as measured through changes in AML Knowledge Questionnaire scores)

OTHER OUTCOMES:
Changes in Attitudes Towards Chemotherapy Scale scores | Day 1. Pre-video screening and post-video
  Changes in Attitudes Towards Chemotherapy Scale scores,
Changes in Decisional Conflict Scale scores | Day 1. Pre-video screening and post-video
  Changes in Decisional Conflict Scale scores
Changes in Anxiety Scores | Day 1. Pre-video screening and post-video
  Changes in Anxiety Scores

CONTACTS AND LOCATIONS:
Overall Officials: Thomas LeBlanc, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hildenbrand JD, Davis DM, El-Jawahri A, Herring KW, Locke SC, Pollak KI, Samsa GP, Steinhauser KE, Troy JD, Ubel PA, Leblanc TW. A novel decision aid for acute myeloid leukemia: a feasibility and preliminary efficacy trial. Support Care Cancer. 2021 Jul;29(7):3563-3569. doi: 10.1007/s00520-020-05864-5. Epub 2020 Nov 6. PMID 33159220